CLINICAL TRIAL: NCT04800068
Title: Expanded Access [Ga-68] PSMA-11 PET Imaging
Status: No longer available | Type: Expanded Access
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Geoffrey Johnson, Principal Investigator, Mayo Clinic
Other Study IDs: 20-013358
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Diagnostic Test: [Ga-68] PSMA-11 PET/CT — Imaging scan
Diagnostic Test: [Ga-68] PSMA-11 PET/MR — Imaging scan

SUMMARY:
In this expanded access IND study, Mayo Clinic in Rochester MN offers [Ga-68] PSMA-11 PET/CT or PET/MR imaging to patients who meet criteria.

DETAILED DESCRIPTION:
[Ga-68] PSMA-11 PET/CT and PET/MR imaging has been shown to allow for accurate detection of metastatic prostate cancer at the time of initial diagnosis and staging of patients with high-risk prostate cancer and at the time of biochemical recurrence. In addition, available data show superiority of metastatic lesion detection with [Ga-68] PSMA-11 PET over conventional imaging. This improved lesion detection has a direct impact on selection of anti-cancer therapy and thus may improve patient outcomes.

Under expanded access IND, enrolled patients will receive a clinical [68Ga] PSMA-11 PET/CT or PET/MR for evaluation of their cancer. Imaging exams must be deemed clinically indicated by a referring provider. Patients will be responsible for the cost of the imaging exam. Access is limited.

ELIGIBILITY:
Participant Groups

There are two participant groups; please refer to the inclusion details below:

Group 1: Untreated High-Risk prostate cancer group (must meet at least one of the following inclusion criteria):

1. Serum prostate-specific antigen (PSA) concentration of 20 ng/mL or more
2. Pathologic criteria of International Society of Uropathology (ISUP) grade group 3-5 (ISUP grades 3-5 are equivalent to pathologic Gleason scores of 4+3, 8, 9 or 10)
3. Local staging of T3 or worse (Indicating that cancer has invaded into tissues outside of the prostate gland, as seen at either CT or MRI)

Biochemically Recurrent prostate cancer group (must meet one of the criteria):

1. In patients who have undergone a prostatectomy, PSA > 0.2 ng/ml on 2 consecutive tests
2. In patients who have undergone definitive prostate radiation, PSA rise ≥ 2 ng/mL above the nadir PSA

Exclusion Criteria: Current exclusion criteria for both groups includes:

1. Patients unable to sign informed consent
2. Patient with a life expectancy less than 6 months
3. Additional exclusion criteria may be added based on demand

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.